CLINICAL TRIAL: NCT05717634
Title: Endometrial Changes in Breast Cancer Women: a Prospective Multicentric Trial.
Brief Title: Endometrial Changes in Breast Cancer Women.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: University of Palermo (Other); University of Padova (Other); Universita di Verona (Other); Federico II University (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); University of Messina (Other); IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Principal Investigator, Benito Chiofalo, MD, PhD, Regina Elena Cancer Institute
Other Study IDs: Regina Elena
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Endometrial Cancer; Endometrial Hyperplasia With Atypia; Breast Cancer; TAM
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia; Breast Neoplasms | interventions — Hysteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TAM: Patients with previous breast cancer with hormonal receptor expression that are treated with tamoxifen.
  Interventions: Diagnostic Test: Hysteroscopy
- Ais: Patients with previous breast cancer with hormonal receptor expression that are treated with Ais.
  Interventions: Diagnostic Test: Hysteroscopy
- No Therapy: Patients with previous breast cancer that are not treated with none hormonal therapies.
  Interventions: Diagnostic Test: Hysteroscopy

INTERVENTIONS:
Diagnostic Test: Hysteroscopy — Patients with suspected endometrial pathology, will undergo hysteroscopy with endometrial biopsy or endometrial lesion excision.
  Other Names: Endometrial biopsy

SUMMARY:
This is a prospective observational multicentric study. The aim is to evaluate the incidence of endometrial cancer and endometrial atypical hyperplasia in patients with previous breast cancer, treated with different adjuvant therapies. The second aim is to identify ultrasonographic soft markers related with endometrial cancer or atipycal hyperplasia.

DETAILED DESCRIPTION:
This is a prospective observational multicentric study. Patient with a history of breast cancer treated with adjuvant hormonal therapies or with no therapies, will be enrolled and followed once a year with physical exam and endovaginal ultrasound. Patients with suspected endometrial pathology will undergo hysteroscopy with endometrial biopsy or endometrial lesion resection.

The aim is to evaluate the incidence of endometrial cancer and endometrial atypical hyperplasia in patients with previous breast cancer, treated with different adjuvant therapies. The second aim is to identify ultrasonographic soft markers related with endometrial cancer or atipycal hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* Personal history of breast cancer

Exclusion Criteria:

* Personal history of other hormonal sensitive cancers
* Assumption of hormones in the previous 5 years
* Previous medical assisted reproduction technique
* Lynch syndrome or BRCA 1/2 mutations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients, divided in three groups: tamoxifen users, aromatase inhibitors users and no therapies.
Sampling Method: Probability Sample
Enrollment: 829 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2023-09-26 (Estimated); Study Completion 2024-01-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of endometrial cancer | One year
  Evaluation of the incidence of endometrial cancer and atypical hyperplasya

SECONDARY OUTCOMES:
Ultrasonographic soft markers of endometrial pathology | One year
  Identification of ultrasonographic soft markers of endometrial pathology

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS "Regina Elena" National Cancer Institute, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-12-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT05717634/Prot_SAP_ICF_000.pdf